CLINICAL TRIAL: NCT01259492
Title: A 40-week, Randomized, Double-blind, Placebo-controlled, Multicenter Efficacy and Safety Study of Methylphenidate HCl Extended Release in the Treatment of Adult Patients With Childhood-onset ADHD
Brief Title: Efficacy and Safety Study of Methylphenidate Hydrochloride Extended Release in Adults With Childhood-onset Attention Deficit/Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CRIT124D2302; 2010-021533-31 (EudraCT Number)
Record Dates: First submitted 2010-12-11; First posted 2010-12-14 (Estimated); Results first posted 2014-04-29 (Estimated); Last update posted 2014-10-07 (Estimated); Status verified 2014-09

CONDITIONS: Attention Deficit/Hyperactivity Disorder
Keywords: Attention Deficit /Hyperactivity Disorder, hyperactivity
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (4):
- Ritalin LA 40 mg (Experimental): In period 1 patients were given Ritalin LA 20 mg and up titrated to 40 mg at week 2, continued in same dose till week 9. Period 2- The dose of study medication was re-titrated for all patients (including those in the Placebo arm during Period 1) starting at 20 mg/day Ritalin LA and increased at weekly intervals in increments of 20 mg/day until reaching the patient's optimal dose 40 mg. Optimal dose was defined as the dose at which the investigator considered an optimal balance between control of symptoms and side effects was maintained for a period of at least one week prior to Week 14. In period 3, patients were re- randomized to either their optimal dose of medication (40, 60, or 80 mg/day) or Placebo from beginning of week 15 to end of week 40.
  Interventions: Drug: Ritalin LA 20 mg
- Ritalin LA 60 mg (Experimental): In period 1 patients were given Ritalin LA 20 mg and up titrated to 40 mg at week 2 and to 60 mg at week 3. Period 2- The dose of study medication was re-titrated for all patients (including those in the Placebo arm during Period 1) starting at 20 mg/day Ritalin LA and increased at weekly intervals in increments of 20 mg/day until reaching the patient's optimal dose 60 mg. Optimal dose was defined as the dose at which the investigator considered an optimal balance between control of symptoms and side effects was maintained for a period of at least one week prior to Week 14.In period 3, patients were re- randomized to either their optimal dose of medication (40, 60, or 80 mg/day) or Placebo from beginning of week 15 to end of week 40.
  Interventions: Drug: Ritalin LA 20 mg; Drug: Ritalin LA 30 mg
- Ritalin LA 80 mg (Experimental): In period 1 patients were given Ritalin LA 20 mg and up titrated to 40 mg at week 2 and to 60 mg at week 3 and to 80 mg at week 4. Period 2- The dose of study medication was re-titrated for all patients (including those in the Placebo arm during Period 1) starting at 20 mg/day Ritalin LA and increased at weekly intervals in increments of 20 mg/day until reaching the patient's optimal dose 60 mg. Optimal dose was defined as the dose at which the investigator considered an optimal balance between control of symptoms and side effects was maintained for a period of at least one week prior to Week 14. In period 3, patients were re- randomized to either their optimal dose of medication (40, 60, or 80 mg/day) or Placebo from beginning of week 15 to end of week 40.
  Interventions: Drug: Ritalin LA 20 mg; Drug: Ritalin LA 30 mg
- Placebo (Placebo Comparator): Period 1- Placebo controlled Period 2 - The dose of study medication was re-titrated for all patients (including those in the Placebo arm during Period 1) starting at 20 mg/day Ritalin LA and increased at weekly intervals in increments of 20 mg/day until reaching the patient's optimal dose (40, 60 or 80 mg). In period 3, patients were re- randomized to either their optimal dose of medication (40, 60, or 80 mg/day) or Placebo from beginning of week 15 to end of week 40.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Placebo Comparator: Placebo
  Arms: Placebo
Drug: Ritalin LA 20 mg — Ritalin LA (a racemic mixture of d- and l-thre-Methylphenidate Hydrochloride (MPH), extended release hard capsules) taken orally once daily in doses of 40, 60, or 80 mg.
  Arms: Ritalin LA 40 mg; Ritalin LA 60 mg; Ritalin LA 80 mg
Drug: Ritalin LA 30 mg — Ritalin LA (a racemic mixture of d- and l-thre-Methylphenidate Hydrochloride (MPH), extended release hard capsules) taken orally once daily in doses of 60, or 80 mg.
  Arms: Ritalin LA 60 mg; Ritalin LA 80 mg

SUMMARY:
This study will evaluate efficacy and safety of methylphenidate hydrochloride extended release compared to placebo in adult patients with childhood-onset attention deficit/hyperactivity disorder (ADHD).

ELIGIBILITY:
Inclusion criteria:

1. Diagnosis of attention deficit/hyperactivity disorder (ADHD) which started in childhood
2. Female patients of childbearing potential must be practicing an acceptable method of contraception.

Exclusion criteria:

1. Patients with body mass index (BMI) less than 18.5 kg/m2 or more than 35 kg/m2
2. History of alcohol or substance abuse within the last six months.
3. History of seizures or use of anticonvulsant medication.
4. Any psychiatric condition that requires medication or may interfere with study participation.
5. Pre-existing cardiovascular disorders including severe hypertension, heart failure, myocardial infraction, etc.
6. Significant respiratory, hepatic, gastrointestinal, renal, hematological or oncologic disorder
7. Diagnosis of glaucoma, hyperthyroidism, pheochromocytoma
8. Diagnosis or family history of Tourette's syndrome
9. Pre-existing cerebrovascular disorders such as cerebral aneurysm, vascular abnormalities including vasculitis or stroke

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 725 (Actual)
Dates: Start 2010-11; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (65):
- United States (19):
  - Novartis Investigative Site, Little Rock, Arkansas
  - Novartis Investigative Site, Beverly Hills, California
  - Novartis Investigative Site, Spring Valley, California
  - Novartis Investigative Site, Bradenton, Florida
  - Novartis Investigative Site, Miami, Florida
  - Novartis Investigative Site, Orlando, Florida
  - Novartis Investigative Site, West Plam Beach, Florida
  - Novartis Investigative Site, Libertyville, Illinois
  - Novartis Investigative Site, Owensboro, Kentucky
  - Novartis Investigative Site, Troy, Michigan
  - Novartis Investigative Site, Las Vegas, Nevada
  - Novartis Investigative Site, Willingboro, New Jersey
  - Novartis Investigative Site, Fargo, North Dakota
  - Novartis Investigative Site, Columbus, Ohio
  - Novartis Investigative Site, Oklahoma City, Oklahoma
  - Novartis Investigative Site, Philadelphia, Pennsylvania
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, Bellevue, Washington
  - Novartis Investigative Site, Seattle, Washington
- Belgium (6):
  - Novartis Investigative Site, Bruges, Belgium
  - Novartis Investigative Site, Heusden-Zolder, Belgium
  - Novartis Investigative Site, Kortenberg, Belgium
  - Novartis Investigative Site, Uccle, Belgium
  - Novartis Investigative Site, Kessel-Lo
  - Novartis Investigative Site, Mechelen
- Colombia (3):
  - Novartis Investigative Site, Santa Fe de Antioquia, Antioquia
  - Novartis Investigative Site, Antioquia
  - Novartis Investigative Site, Bogotá
- Novartis Investigative Site, Århus C, Denmark
- Germany (27):
  - Novartis Investigative Site, Ahrensburg, Germany
  - Novartis Investigative Site, Bamberg, Germany
  - Novartis Investigative Site, Berlin, Germany
  - Novartis Investigative Site, Essen, Germany
  - Novartis Investigative Site, Hamburg, Germany
  - Novartis Investigative Site, Kiel, Germany
  - Novartis Investigative Site, Ludwigsburg, Germany
  - Novartis Investigative Site, Mainz, Germany
  - Novartis Investigative Site, München, Germany
  - Novartis Investigative Site, Naumburg, Germany
  - Novartis Investigative Site, Nuremberg, Germany
  - Novartis Investigative Site, Wolfsburg, Germany
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Ellwangen
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Hagen
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Homburg
  - Novartis Investigative Site, Landau
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Limburg
  - Novartis Investigative Site, Mannheim
  - Novartis Investigative Site, Siegen
  - Novartis Investigative Site, Ulm
  - Novartis Investigative Site, Westerstede/Oldenburg
  - Novartis Investigative Site, Würzburg
- Norway (2):
  - Novartis Investigative Site, Porsgrunn, Norway
  - Novartis Investigative Site, Skien
- Novartis Investigative Site, Singapore, Singapore
- South Africa (3):
  - Novartis Investigative Site, Benoni
  - Novartis Investigative Site, Melrose Arch
  - Novartis Investigative Site, Pretoria
- Sweden (3):
  - Novartis Investigative Site, Luleå
  - Novartis Investigative Site, Malmo
  - Novartis Investigative Site, Stockholm

REFERENCES:
- [Derived] Huss M, Ginsberg Y, Tvedten T, Arngrim T, Philipsen A, Carter K, Chen CW, Kumar V. Methylphenidate hydrochloride modified-release in adults with attention deficit hyperactivity disorder: a randomized double-blind placebo-controlled trial. Adv Ther. 2014 Jan;31(1):44-65. doi: 10.1007/s12325-013-0085-5. Epub 2013 Dec 27. PMID 24371021

RESULTS

PARTICIPANT FLOW:
Period: Period 1 (9 Weeks)
Arm/Group | Ritalin LA 40 mg | Ritalin LA 60 mg | Ritalin LA 80 mg | Placebo
Started | 181 | 182 | 181 | 181
Full Analysis Set | 174 | 175 | 179 | 172
Completed | 152 ("Completed" indicates patients entered Period 2.) | 141 (Completed = entered Period 2) | 138 (Completed = entered Period 2) | 153 (Completed = entered Period 2)
Not Completed | 29 | 41 | 43 | 28
Not completed — Adverse Event | 13 | 18 | 26 | 3
Not completed — Lack of Efficacy | 2 | 2 | 4 | 11
Not completed — Withdrawal by Subject | 5 | 8 | 6 | 7
Not completed — Lost to Follow-up | 4 | 6 | 3 | 4
Not completed — Administrative Problems | 0 | 1 | 1 | 2
Not completed — Protocol Violation | 5 | 6 | 3 | 1
Period: Period 2 (Week 10 to Week 14)
Arm/Group | Ritalin LA 40 mg | Ritalin LA 60 mg | Ritalin LA 80 mg | Placebo
Started | 152 (Treatment arms including Placebo indicate patients belong to respective treatment arms in Period 1) | 141 | 138 | 153
Completed | 127 (Completed = entered Period 3) | 123 (Completed = entered Period 3) | 114 (Completed = entered Period 3) | 125 (Completed = entered Period 3)
Not Completed | 25 | 18 | 24 | 28
Not completed — Adverse Event | 3 | 4 | 7 | 8
Not completed — Lack of Efficacy | 13 | 7 | 7 | 13
Not completed — Withdrawal by Subject | 6 | 2 | 8 | 4
Not completed — Lost to Follow-up | 3 | 3 | 1 | 3
Not completed — Protocol Violation | 0 | 2 | 1 | 0
Period: Period 3 (Week 15 to End of Week 40)
Arm/Group | Ritalin LA 40 mg | Ritalin LA 60 mg | Ritalin LA 80 mg | Placebo
Started | 114 (In period 3, all 489 patients who completed period 2 were re-randomized to 4 arms.) | 132 | 120 | 123
Full Analysis Set | 110 | 128 | 114 | 115
Completed | 60 (completed study) | 63 (completed study) | 70 (completed study) | 42 (completed study)
Not Completed | 54 | 69 | 50 | 81
Not completed — Adverse Event | 5 | 11 | 6 | 5
Not completed — Abnormal Lab value(s) | 0 | 0 | 0 | 1
Not completed — Abnormal Test Procedure Result(s) | 0 | 0 | 1 | 0
Not completed — Lack of Efficacy | 28 | 42 | 29 | 62
Not completed — Patient no longer requires study drug | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 12 | 6 | 4 | 3
Not completed — Lost to Follow-up | 3 | 4 | 6 | 3
Not completed — Administrative Problems | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 5 | 6 | 3 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ritalin LA 40 mg | Ritalin LA 60 mg | Ritalin LA 80 mg | Placebo | Total
Number analyzed (Participants) | 181 | 182 | 181 | 181 | 725
Age, Customized [Number; unit: Participants] — Period 1
  Participants
    18-30 | 72 | 78 | 71 | 66 | 287
    31-40 | 39 | 45 | 40 | 38 | 162
    41-50 | 56 | 45 | 57 | 47 | 205
    51-60 | 14 | 14 | 13 | 30 | 71
Age, Customized [Number; unit: Participants] — Period 3
  Participants
    18-30 | 53 | 46 | 34 | 52 | 185
    31-40 | 19 | 32 | 27 | 27 | 105
    41-50 | 32 | 41 | 45 | 31 | 149
    51-60 | 10 | 13 | 14 | 13 | 50
Sex: Female, Male [Count of Participants; unit: Participants] — Period 1
  Participants
    Female | 87 | 77 | 86 | 80 | 330
    Male | 94 | 105 | 95 | 101 | 395
Gender [Number; unit: Participants] — Period 3
  Participants
    Female | 60 | 58 | 46 | 52 | 216
    Male | 54 | 74 | 74 | 71 | 273

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline of Period 1 (Baseline 1) to End of Period 1 on Attention-Deficit/Hyperactivity Disorder Rating Scale (DSM-IV ADHD RS) Total Score by Treatment
Description: Attention-Deficit/Hyperactivity Disorder Rating Scale (DSM-IV ADHD RS) total score consists of 18 items directly adapted from the ADHD symptom list according to the DSM-IV. The DSM-IV ADHD RS total score was calculated as the sum of the Inattentive and the Hyperactive-Impulsive subscores. The 18 items are rated from 0 ("Never") to 4 ("Very often"). The total score ranges from 0(least symptomatic) to 72 (most symptomatic). Decrease in the DSM-IV ADHD RS total score indicates improvement, therefore a greater decrease (change at Final Visit compared to baseline) indicates a greater improvement in ADHD symptoms. 30% improvement: 100×(DSM-IV ADHD RS total score during Period 1 - DSM-IV ADHD RS total score at randomization(visit 2))/DSM-IV ADHD RS total score at randomization (visit 2) <= - 30%.
Time Frame: Baseline 1 to End of Period 1 (Week 9)
Population: Full Analysis Set for Period 1 (FAS P1) - all randomized patients who take one dose of study medication in period 1. Patients will be assigned to their randomized fixed dose. Patients with both baseline and post-baseline (end of week 9) assessments were included.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Ritalin LA 40 mg | Ritalin LA 60 mg | Ritalin LA 80 mg | Placebo
Number analyzed (Participants) | 160 | 155 | 156 | 161
Units on a Scale | 16.0 (12.18) | 14.7 (10.12) | 16.8 (11.36) | 9.7 (11.05)

2. Primary Outcome: Change From Baseline Period 1 (Baseline 1) to End of Period 1 on Sheehan Disability Scale (SDS) Total Score by Treatment
Description: SDS, a 5-self-rated questionnaire to measure the extent a pt's disability due to an illness/health problem interferes with work/school, social life/leisure, family life/home. First 3 items, pts are asked how their symptoms disrupted their reg. activities over the past 7d in ea. using a scale from 0(not at all)-10(extremely) Ea. subscale(work disability, social life disability, family life disability) can be scored independently or combined into a total score(sum of the non-missing responses for items 1-3)from 0-30,higher scores indicate significant functional impairmt. Subscale scores >5 suggest impairment in that subscale area. Final 2 items ask pts about the # of days their symptoms caused them to miss school/work and # of days their symptoms caused them to be underproductive at school/work.(These items were not included in the total score.) Before responding to SDS items 1-3, pts were verbally instructed to recall the past 7d, items 4-5 refer to the last week w/in the item wording.
Time Frame: Baseline 1 to End of Period 1 (Week 9)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Ritalin LA 40 mg | Ritalin LA 60 mg | Ritalin LA 80 mg | Placebo
Number analyzed (Participants) | 151 | 146 | 148 | 152
Units on a Scale | 6.4 (7.54) | 4.7 (7.08) | 6.1 (7.31) | 2.9 (7.47)

3. Primary Outcome: Percentage of Participants With Treatment Failures During Period 3
Description: Treatment failure is defined as: 100×(DSM-IV ADHD RS total score during Period 3 - DSM-IV ADHD RS total score at re-randomization (visit 13))/DSM-IV ADHD RS total score at re-randomization (visit 13) >= 30% AND 100×(DSM-IV ADHD RS total score during Period 3 - DSM-IV ADHD RS total score at randomization (visit 2))/DSM-IV ADHD RS total score at randomization (visit 2) > - 30%. The ADHD-RS-IV is an 180item clinician rated scale to assess ADHD by DSM-IV-TR, defined criteria using symptom terminology appropriate for the adult population. Each item pertains to inattention (odd-numbered) or hyperactivity/impulsivity (even-numbered) and is scored on a scale of 0 (no symptoms) to 3 (severe symptoms). A total added score can range from 0-54
Time Frame: Baseline Period 1 (Baseline 1) and Baseline Period 3 (Baseline 2) to End of Week 40
Population: Full Analysis Set for Period 3 (FAS P3) - all re-randomized patients who take one dose of study medication in period 3. One patient in Ritalin LA 80mg did not have post baseline 2 measurements and was not included in the categories under without imputation.
Measure: Number; unit: Percentage of participants
Arm/Group | Ritalin LA 40 mg | Ritalin LA 60 mg | Ritalin LA 80 mg | Placebo
Number analyzed (Participants) | 110 | 128 | 114 | 115
Percentage of participants
  Without Imputation - Treatment failure | 11.8 (7.54) | 20.3 (7.08) | 17.5 (7.31) | 43.5 (7.47)
  Without Imputation - Not treatment failure | 54.5 | 50.0 | 56.1 | 31.3
  Without Imputation missing failure status | 33.6 | 29.7 | 25.4 | 25.2
  With Imputation - Treatment failure | 16.4 | 26.6 | 20.2 | 49.6
  With Imputation - Not treatment failure | 83.6 | 73.4 | 79.8 | 50.4

4. Secondary Outcome: Percentage of Patients With Improvement on Clinical Global Impression - Improvement Scale (CGI-I) From Baseline Period 1 (Baseline 1) to End of Period 1
Description: On the CGI-I scale, a lower score reflects greater improvement between 1 and 3, a score of 4 is "no change", scores higher than 4 reflect worsening. The CGI-I consists of 7 ratings that range from 1 = "Very much improved" to 7 ="Very much worse". Improvement on the CGI-I scale is defined as a visit rating of 1 "very much improved" or 2 "much improved" on the CGI-I scale. Percentage has been calculated from the evaluable patients (N) as Percentage = n/N * 100.
Time Frame: Baseline 1 to End of Period 1 (Week 9)
Population: Full Analysis Set for Period 1 (FAS P1) - all randomized patients who take one dose of study medication in period 1. Patients will be assigned to their randomized fixed dose. Evaluable patients with both baseline and post-baseline (end of week 9) assessments were included.
Measure: Number; unit: Percentage of Patients
Arm/Group | Ritalin LA 40 mg | Ritalin LA 60 mg | Ritalin LA 80 mg | Placebo
Number analyzed (Participants) | 160 | 155 | 156 | 161
Percentage of Patients | 56.3 | 54.8 | 57.1 | 31.7

5. Secondary Outcome: Change From Baseline 1 in DSM-IVADHD RS Total Score, SDS Total Score, The Conners' Adult ADHD Rating Scale Observer Short Version (CAARS-O:S) Total Score and Adult Self-Report Scale (ASRS) Total Score at the End of Period 2 (Visit 13/ Week 14)
Description: DSM-IV ADHD RS consists of 18 items directly adapted from the ADHD symptom list according to the DSM-IV. The SDS is a five-item, self-rated questionnaire that has been used widely in clinical trials and observational studies. CAARS-O: S consists of 26 items and 6 subscales: Inattention/Memory Problems, Hyperactivity/Restlessness, Impulsivity/Emotional Lability, Problems with Self-Concept, ADHD Index, and Inconsistency Index and is rated by someone close to the patient in their daily life such as a spouse, friend, or coworker. The Adult Self-Report Scale (ASRS) is a self-rating scale designed to assess Attention-Deficit/Hyperactivity Disorder (ADHD) symptoms. The 18 items are written to reflect the DSM-IV diagnostic criteria for ADHD and are rated from 0 ("Never") to 4 ("Very often").
Time Frame: Baseline 1 to End of Period 2 (Week 14)
Population: Full Analysis Set for Period 2 (FAS P2) - all randomized patients who took one dose of study medication in Period 2
Measure: Mean (Standard Deviation); unit: Score on Scale
Groups:
- ALL Ritalin LA Group: This group combined all Ritalin patients on 40 mg, 60 mg and 80 mg. n=492
Arm/Group | ALL Ritalin LA Group
Number analyzed (Participants) | 563
Score on Scale
  DSM-IV ADHD RS total score n=494 | 24.8 (8.97)
  SDS total score n=480 | 10.1 (7.25)
  CAARS-O:S total score n=411 | 15.5 (15.25)
  ASRS total score n=490 | 23.2 (14.16)

6. Secondary Outcome: Number of Participants With Clinical Global Impression - Improvement Scale (CGI-I) Rating at the End of Period 2 (Visit 13/ Week 14)
Description: CGI-I assesses the overall change of illness relative to baseline. CGI-I consists of 7 ratings that range from 1 = "very much improved", 2 = "much improved", 3 = "minimally improved", 4 = "no change from baseline", 5 = "minimally worse", 6 = "much worse" 7 = "very much worse"
Time Frame: Baseline 1 to End of Period 2 (Week 14)
Population: Full Analysis Set for Period 2 (FAS P2) - all randomized patients who took one dose of study medication in Period 2 Patients with CGI-I assessment both at Baseline 1 and Period 2 was included.
Measure: Number; unit: number of participants
Arm/Group | ALL Ritalin LA Group
Number analyzed (Participants) | 563
number of participants
  very much improved | 195
  much improved | 230
  minimally improved | 42
  no change | 16
  minimally worse | 7
  much worse | 2
  very much worse | 0

7. Secondary Outcome: Number of Participants With Clinical Global Impression - Improvement Scale Severity of Illness (CGI-S) Rating at the End of Period 2 (Visit 13/ Week 14)
Description: CGI-S assesses the patient's current illness state. CGI-S consists of 7 ratings that range from 1 = "normal, not at all ill" , 2 = "borderline mentally ill", 3 =" mildly ill", 4 = "moderately ill", 5 = "markedly ill", 6 = "severely ill", 7 = "among the most extremely ill patients"
Time Frame: Baseline 1 to End of Period 2 (Week 14)
Population: Full Analysis Set for Period 2 (FAS P2) - all randomized patients who took one dose of study medication in Period 2; Patients with CGI-S assessment both at Baseline 1 and Period 2 was included.
Measure: Number; unit: number of participants
Arm/Group | ALL Ritalin LA Group
Number analyzed (Participants) | 563
number of participants
  Normal, not ill at all | 91
  borderline mentally ill | 151
  mildly ill | 193
  moderately ill | 50
  markedly ill | 7
  severely ill | 0
  among the most extremely ill patients | 0

8. Secondary Outcome: Change From Baseline Period 3 (Baseline 2) to End of Period 3 on DSM-IV Attention-Deficit/Hyperactivity Disorder Rating Scale ADHD RS Total Score by Treatment
Description: The ADHD-RS-IV is an 180 item clinician rated scale to assess ADHD by DSM-IV-TR, defined criteria using symptom terminology appropriate for the adult population. Each item pertains to inattention (odd-numbered) or hyperactivity/impulsivity (even-numbered) and is scored on a scale of 0 (no symptoms) to 3 (severe symptoms). A total added score can range from 0-54.
Time Frame: Baseline 2 to end of Period 3 (end of withdrawal period 40 weeks)
Population: Full Analysis Set for Period 3 (FAS P3) - all re-randomized patients who take one dose of study medication in period 3. Patients will be assigned to their re-randomized treatment; Ritalin (pooled doses) or placebo.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Ritalin LA 40 mg | Ritalin LA 60 mg | Ritalin LA 80 mg | Placebo
Number analyzed (Participants) | 101 | 121 | 106 | 106
Units on a Scale | 3.0 (10.07) | 5.1 (10.85) | 2.6 (8.67) | 9.3 (11.95)

9. Secondary Outcome: Change From Baseline Period 3 (Baseline 2) to End of Period 3 on SDS Total Score by Treatment
Description: The Sheehan Disability Scale (SDS) is a self-rating scale designed to assess the extent to which the patient's work social life/leisure activities and home life are impaired by his or her symptoms. The scale generates 4 scores: a work disability score, a social life disability score, a family life disability score and a total score. To get a total score the 3 individual scores (work: social life: family life) are totaled. The maximum possible score is 30 The higher the score, the more "impaired" a patient's work, social life, family life is.
Time Frame: Baseline 2 to end of Period 3 (end of withdrawal period 40 weeks)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Ritalin LA 40 mg | Ritalin LA 60 mg | Ritalin LA 80 mg | Placebo
Number analyzed (Participants) | 100 | 118 | 101 | 102
Units on a Scale | 2.1 (6.34) | 2.3 (7.19) | 2.0 (6.81) | 5.0 (8.15)

10. Secondary Outcome: Number of Patients With Worsening on CGI-I Scale From Baseline Period 3 (Baseline 2) to End of Period 3 by Treatment
Description: On the CGI-I scale, a lower score reflects greater improvement between 1 and 3, a score of 4 is "no change", scores higher than 4 reflect worsening. The CGI-I consists of 7 ratings that range from 1 = "Very much improved" to 7 ="Very much worse". Improvement on the CGI-I scale is defined as a visit rating of 1 "very much improved" or 2 "much improved" on the CGI-I scale.
Time Frame: Baseline 2 to end of Period 3 (end of withdrawal period 40 weeks)
Population: Full Analysis Set for Period 3 (FAS P3) - all re-randomized patients who take one dose of study medication in period 3. Patients will be assigned to their re-randomized treatment; Ritalin (pooled doses) or placebo. Evaluable patients with both baseline 2 and post-baseline (end of week 40) assessments were included.
Measure: Number; unit: participants
Arm/Group | Ritalin LA 40 mg | Ritalin LA 60 mg | Ritalin LA 80 mg | Placebo
Number analyzed (Participants) | 102 | 120 | 108 | 108
participants | 6 | 13 | 5 | 21

11. Secondary Outcome: Number of Patients With Worsening on CGI-S Scale From Baseline Period 3 (Baseline 2) to End of Period 3 by Treatment
Description: as for outcome 7
Time Frame: Baseline 2 to end of Period 3 (end of withdrawal period 40 weeks)
Population: as for outcome 10
Measure: Number; unit: Participants
Arm/Group | Ritalin LA 40 mg | Ritalin LA 60 mg | Ritalin LA 80 mg | Placebo
Number analyzed (Participants) | 102 | 120 | 107 | 110
Participants | 39 | 50 | 35 | 72

12. Secondary Outcome: Change From Baseline Period 3 (Baseline 2) to End of Period 3 in Conners Adult ADHD Rating Scales Observer: Short Version (CAARS-O:S:) Total Score by Treatment
Description: CAARS is an instrument to assess ADHD symptoms and behaviors in adults. This study utilizes the Observer Short Version (CAARS-O: S), consisting of 26 items and 6 subscales: Inattention/Memory Problems, Hyperactivity/Restlessness, Impulsivity/Emotional Lability, Problems with Self-Concept, ADHD Index (to distinguish ADHD adults from non-clinical adults), and Inconsistency Index (to identify random or careless responding) and is rated by someone close to the patient in their daily life such as a spouse, friend, or coworker. The observer is asked to notice the patient carefully and decide how much or how frequently each of the 26 items of the scale describes the patient recently. The response to every question in increasing order of severity is "not at all, never = 0; Just a little, once in a while = 1; Pretty much, often = 2; Very much, very frequently = 3". The total score combined from all the 26 items ranges from 0 to 88.
Time Frame: Baseline 2 to end of Period 3 (end of withdrawal period 40 weeks)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Ritalin LA 40 mg | Ritalin LA 60 mg | Ritalin LA 80 mg | Placebo
Number analyzed (Participants) | 76 | 92 | 83 | 78
Units on a scale | -2.7 (11.74) | 1.7 (12.00) | -0.2 (14.23) | 2.9 (15.26)

13. Secondary Outcome: Change From Baseline Period 3 (Baseline 2) to End of Period 3 in ASRS Total Score by Treatment
Description: The ASRS is a self-rating scale designed to assess ADHD symptoms in adults and is now part of the World Health Organization Composite International Diagnostic Interview. It consists of 18 items written to reflect the DSM-IV diagnostic criteria for ADHD and are rated from 0 ("Never") to 4 ("Very often"). The total score ranges from 0 to 72.
Time Frame: Baseline 2 to end of Period 3 (end of withdrawal period 40 weeks)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Ritalin LA 40 mg | Ritalin LA 60 mg | Ritalin LA 80 mg | Placebo
Number analyzed (Participants) | 99 | 119 | 105 | 103
Units on a scale | 3.0 (12.64) | 3.8 (12.66) | 3.0 (11.54) | 8.0 (16.39)

ADVERSE EVENTS:
Description: N of safety analysis set for Period 1=722. Data in the entire three periods were included. A patient may be counted under both treatment arms. Which means, if a patient received placebo in Period 1 and Ritalin in Period 3, he/she was counted under both 695 and 275. That is why 695+275 > 722.
Groups:
- All Ritalin LA: All Ritalin LA:
  In period 1 patients were given Ritalin LA 20 mg and up titrated to 40 mg at week 2 and to 60 mg at week 3 and to 80 mg at week 4. Period 2- The dose of study medication was re-titrated for all patients (including those in the Placebo arm during Period 1) starting at 20 mg/day Ritalin LA and increased at weekly intervals in increments of 20 mg/day until reaching the patient's optimal dose 60 mg. Optimal dose was defined as the dose at which the investigator considered an optimal balance between control of symptoms and side effects was maintained for a period of at least one week prior to Week 14. In period 3, patients continued on their optimal dose.
Arm/Group | All Ritalin LA | Placebo
Serious Adverse Events (participants affected / at risk) | 9/695 | 4/275
Other Adverse Events (participants affected / at risk) | 517/695 | 104/275
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Ritalin LA (N=695) | Placebo (N=275)
Sudden hearing loss (Ear and labyrinth disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
Goitre (Endocrine disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Eye infection (Infections and infestations) | 0 | 1
Infected bites (Infections and infestations) | 1 | 0
Localised infection (Infections and infestations) | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Adjustment disorder (Psychiatric disorders) | 1 | 0
Agitation (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Panic attack (Psychiatric disorders) | 1 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Ovarian cyst ruptured (Reproductive system and breast disorders) | 1 | 0
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Ritalin LA (N=695) | Placebo (N=275)
Palpitations (Cardiac disorders) | 63 | 2
Tachycardia (Cardiac disorders) | 56 | 0
Vertigo (Ear and labyrinth disorders) | 18 | 2
Abdominal pain upper (Gastrointestinal disorders) | 29 | 8
Diarrhoea (Gastrointestinal disorders) | 31 | 14
Dry mouth (Gastrointestinal disorders) | 142 | 4
Nausea (Gastrointestinal disorders) | 93 | 9
Fatigue (General disorders) | 64 | 14
Feeling jittery (General disorders) | 15 | 0
Irritability (General disorders) | 50 | 9
Thirst (General disorders) | 15 | 1
Influenza (Infections and infestations) | 15 | 5
Nasopharyngitis (Infections and infestations) | 122 | 22
Sinusitis (Infections and infestations) | 15 | 2
Upper respiratory tract infection (Infections and infestations) | 17 | 9
Blood pressure increased (Investigations) | 22 | 3
Weight decreased (Investigations) | 27 | 2
Decreased appetite (Metabolism and nutrition disorders) | 182 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 27 | 8
Dizziness (Nervous system disorders) | 55 | 5
Headache (Nervous system disorders) | 178 | 39
Somnolence (Nervous system disorders) | 8 | 6
Tremor (Nervous system disorders) | 31 | 1
Agitation (Psychiatric disorders) | 23 | 0
Anxiety (Psychiatric disorders) | 50 | 3
Depressed mood (Psychiatric disorders) | 20 | 4
Depression (Psychiatric disorders) | 20 | 1
Initial insomnia (Psychiatric disorders) | 34 | 2
Insomnia (Psychiatric disorders) | 77 | 9
Nervousness (Psychiatric disorders) | 30 | 0
Restlessness (Psychiatric disorders) | 48 | 7
Sleep disorder (Psychiatric disorders) | 28 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 22 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 16 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 62 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigators are NOT employed by the organization sponsoring the study. Other disclosure agreement that restricts the right of the PI to discuss or publish trial results after the trial is completed. The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial.